CLINICAL TRIAL: NCT01401530
Title: Phase1/1b Clinical Trial of E7777 for the Treatment of Patients With Peripheral T-Cell Lymphoma
Brief Title: E7777 for the Treatment of Patients With Peripheral T-Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7777-J081-101
Record Dates: First submitted 2011-07-18; First posted 2011-07-25 (Estimated); Results first posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-04

CONDITIONS: Peripheral T-Cell Lymphoma
Keywords: Neoplasms; Neoplasms by Histologic Type; Lymphoma; Non-Hodgkin; T- Cell; Lymphatic Diseases; Lymphoproliferative Disorders; lmmune System Diseases; lmmunoproliferative Disorders
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Neoplasms; Neoplasms by Histologic Type; Lymphoma; Lymphatic Diseases; Lymphoproliferative Disorders | interventions — denileukin diftitox

ARMS (1):
- E7777 (Experimental)
  Interventions: Biological: denileukin diftitox (E7777)

INTERVENTIONS:
Biological: denileukin diftitox (E7777) — E7777 will be administered by intravenous (IV) infusion for 5 days from Day 1 through 5 of each cycle (21 days/cycle) with 8 cycles in maximum for E7777 alone therapy. E7777 dose will be escalated from 6 micro-g/kg/day to 12, 15 and then to 18 in a stepwise fashion.

SUMMARY:
The purpose of this Phase 1 study is to determine the maximum tolerated dose (MTD) through observation of dose limiting toxicity (DLT), which is in advance defined, in patients with peripheral or cutaneous T-cell lymphoma.

ELIGIBILITY:
lnclusion Criteria:

* Male and female patients 20 to less than 80 years of age at the time of informed consent
* Patients histologically or cytologically diagnosed to have peripheral T -cell lymphoma
* Patients with a history of chemotherapy (including PUVA and retinoid) that resulted in relapse, recurrence and treatment resistance (just for the administration of E7777 alone)
* Patients subject to CHOP therapy and without a history of prior treatment with anthracycline or anthraquinone anticancer drugs (just for the administration of E7777 in combination with CHOP therapy)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
* No carry-over of beneficial or adverse effects of the prior treatment that may affect the safety evaluation of the investigational drug (excluding Grade 1 neuropathy and alopecia)

Exclusion Criteria:

* Brain metastasis with clinical symptoms which requires treatment
* Serious systemic infection requiring intensive treatment
* Serious complications or histories
* History of hypersensitivity to protein therapeutics
* Known to be positive for HIV antibody, HCV antibody, or HBs antigen
* History of malignancy other than peripheral T-cell lymphoma and less than five years have elapsed since the last remission
* Patients who have undergone allogeneic hematopoietic stem cell transplantation
* Patients with a relapse within 6 months after autologous hematopoietic stem-cell transplantation

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-07; Primary Completion 2015-08 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tadashi Nakanishi, Study Director — Eisai Co., Ltd.
Locations (4):
- Japan (4):
  - Nagoya, Aichi-ken
  - Kashiwa, Chiba
  - Isehara, Kanagawa
  - Chuo-ku, Tokyo

REFERENCES:
- [Derived] Ohmachi K, Ando K, Ogura M, Uchida T, Tobinai K, Maruyama D, Namiki M, Nakanishi T. E7777 in Japanese patients with relapsed/refractory peripheral and cutaneous T-cell lymphoma: A phase I study. Cancer Sci. 2018 Mar;109(3):794-802. doi: 10.1111/cas.13513. Epub 2018 Feb 26. PMID 29363235

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: 6 ug/kg/Day Denileukin Diftitox: Denileukin diftitox was intravenously (IV) infused for 60 minutes (±10 minutes) daily from Day 1 through Day 5 of each Cycle (1 cycle = 3 weeks).
- Cohort 2: 9 ug/kg/Day Denileukin Diftitox; Cohort 3: 12 ug/kg/Day Denileukin Diftitox: Denileukin diftitox was IV-infused for 60 minutes (±10 minutes) daily from Day 1 through Day 5 of each Cycle (1 cycle = 3 weeks).
Period: Overall Study
Arm/Group | Cohort 1: 6 ug/kg/Day Denileukin Diftitox | Cohort 2: 9 ug/kg/Day Denileukin Diftitox | Cohort 3: 12 ug/kg/Day Denileukin Diftitox
Started | 3 | 7 | 3
Completed | 0 | 1 | 0
Not Completed | 3 | 6 | 3
Not completed — Disease Progression | 1 | 2 | 1
Not completed — Adverse Event | 1 | 1 | 1
Not completed — Participant Choice | 1 | 2 | 1
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least one dose of the study drug with at least one evaluable, post-baseline safety datum.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: 6 ug/kg/Day Denileukin Diftitox | Cohort 2: 9 ug/kg/Day Denileukin Diftitox | Cohort 3: 12 ug/kg/Day Denileukin Diftitox | Total
Number analyzed (Participants) | 3 | 7 | 3 | 13
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.7 (5.51) | 49.9 (17.74) | 66.3 (4.16) | 58.2 (15.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 1 | 5
  Male | 2 | 4 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) and Recommended Dose (RD)
Description: The MTD was defined as the maximum tolerated dose observed after the evaluation of dose limiting toxicity (DLT) in Cycle 1 with 6 participants. If it was judged that the dose was not tolerated and DLT was confirmed in only 3 participants in the lower dose cohort, 3 other participants were to be added and tolerability was evaluated with 6 participants in total. The RD was to be comprehensively determined based on the MTD and safety data. Participants not evaluable for DLT were defined as participants found to be ineligible or in whom DLT evaluation was impossible due to premature termination for reasons other than toxicities in the judgement of the Sponsor, among those who had received at least one dose of the investigational drug after enrollment.
Time Frame: For each dose, first dose of study drug (Cycle 1 Day 1) to end of Cycle 1 (Day 21) (1 cycle = 3 weeks)
Population: DLT evaluation analysis set included all participants after excluding, from the Safety Analysis Set, participants who were non-evaluable for DLT.
Measure: Number; unit: ug/kg/day
Groups:
- Denileukin Diftitox: Denileukin diftitox was intravenously (IV) infused for 60 minutes (±10 minutes) daily from Day 1 through Day 5 of each Cycle (1 cycle = 3 weeks).
Arm/Group | Denileukin Diftitox
Number analyzed (Participants) | 12
ug/kg/day | 9

2. Secondary Outcome: Number of Participants With Non-Serious Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) as a Measure of Safety and Tolerability of Denileukin Diftitox
Description: Safety assessments consisted of monitoring and recording all AEs and SAEs; regular monitoring of hematology, blood coagulation, blood chemistry, and urinalysis values; periodic measurement of vital signs, body weight, 12-lead electrocardiograms (ECGs), Eastern Cooperative Oncology Group performance status, physical examination findings, and ophthalmological examination findings. TEAEs were defined as an AE that had an onset date, or worsening in severity from baseline (pre-treatment), on or after the first dose of study drug up to the last assessment. Treatment-related TEAEs included TEAEs that were considered by the investigator to be possibly or probably related to study drug. SAEs were defined as any untoward medical occurrence which results in death, was life-threatening, required hospitalization or prolonged hospitalization, resulted in persistent or significant disability/incapacity, or caused a congenital anomaly/birth defect.
Time Frame: From date of first dose up to 30 days after the last dose of study treatment, up to approximately 4 years 2 months
Population: Safety Analysis Set (SAS) included all participants who received at least one dose of the study drug with at least one evaluable, post-baseline safety datum.
Measure: Number; unit: Participants
Groups:
- Cohort 1: 6 ug/kg/Day Denileukin Diftitox: Denileukin diftitox (6 ug/kg/day) was IV-infused for 60 minutes (±10 minutes) daily from Day 1 through Day 5 of each Cycle (1 cycle = 3 weeks).
- Cohort 2: 9 ug/kg/Day Denileukin Diftitox: Denileukin diftitox (9 ug/kg/day) was IV-infused for 60 minutes (±10 minutes) daily from Day 1 through Day 5 of each Cycle (1 cycle = 3 weeks).
- Cohort 3: 12 ug/kg/Day Denileukin Diftitox: Denileukin diftitox (12 ug/kg/day) was IV-infused for 60 minutes (±10 minutes) daily from Day 1 through Day 5 of each Cycle (1 cycle = 3 weeks).
Arm/Group | Cohort 1: 6 ug/kg/Day Denileukin Diftitox | Cohort 2: 9 ug/kg/Day Denileukin Diftitox | Cohort 3: 12 ug/kg/Day Denileukin Diftitox
Number analyzed (Participants) | 3 | 7 | 3
Participants
  TEAEs | 3 | 7 | 3
  Treatment-related TEAEs | 3 | 7 | 3
  Treatment-emergent SAEs | 1 | 3 | 1
  Death | 0 | 0 | 1

3. Secondary Outcome: Maximum Serum Concentration (Cmax) of Denileukin Diftitox
Description: Cmax was defined as the maximum observed concentration of denileukin diftitox following administration of study treatment on Cycle 1 Day 1 and was obtained directly from the measured serum concentration-time curves. Blood samples were collected before and 30 minutes after the start of infusion and immediately (0 minutes), 30, 60, 90, and 120 minutes after the end of infusion of denileukin diftitox. The samples were analyzed for the amount of denileukin diftitox in the serum using a validated ligand-binding assay with a lower limit of quantitation (LLOQ) of 30 nanograms per milliliter (ng/mL). Serum pharmacokinetic (PK) data were analyzed using a non-compartmental analysis approach to obtain individual participant estimates of Cmax, which was then summarized as the median and full range for all participants and expressed as ng/mL.
Time Frame: Cycle 1 (Day 1)
Population: PK analysis set included all participants in whom at least one PK parameter could be calculated.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cohort 1: 6 ug/kg/Day Denileukin Diftitox | Cohort 2: 9 ug/kg/Day Denileukin Diftitox | Cohort 3: 12 ug/kg/Day Denileukin Diftitox
Number analyzed (Participants) | 3 | 5 | 2
ng/mL | 129 [101 to 130] | 149 [135 to 245] | 181 [158 to 204]

4. Secondary Outcome: Time to Cmax (Tmax) of Denileukin Diftitox in Serum
Description: Blood samples were collected before and 30 minutes after the start of infusion and immediately (0 minutes), 30, 60, 90, and 120 minutes after the end of infusion of denileukin diftitox. The samples were analyzed for the amount of denileukin diftitox in the serum using a validated ligand-binding assay with a LLOQ of 30 ng/mL. Serum PK data were analyzed using a non-compartmental analysis approach to obtain individual participant estimates of Tmax, which was then summarized as the median and full range for all participants and expressed in minutes.
Time Frame: Cycle 1 (Day 1)
Population: PK analysis set
Measure: Median (Full Range); unit: Minutes
Arm/Group | Cohort 1: 6 ug/kg/Day Denileukin Diftitox | Cohort 2: 9 ug/kg/Day Denileukin Diftitox | Cohort 3: 12 ug/kg/Day Denileukin Diftitox
Number analyzed (Participants) | 3 | 5 | 2
Minutes | 64.000 [64.00 to 86.00] | 64.000 [60.00 to 98.00] | 74.500 [64.00 to 85.00]

5. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time 0 to Time of Last Quantifiable Concentration (AUC(0-t))
Description: Blood samples were collected before and 30 minutes after the start of infusion and immediately (0 minutes), 30, 60, 90, and 120 minutes after the end of infusion of denileukin diftitox. The samples were analyzed for the amount of denileukin diftitox in the serum using a validated ligand-binding assay with a LLOQ of 30 ng/mL. Serum PK data were analyzed using a non-compartmental analysis approach to obtain individual participant estimates of AUC(0-t), which was then summarized as the median and full range for all participants and expressed as nanograms*minutes per milliliter (ng*min/mL).
Time Frame: Cycle 1 (Day 1)
Population: PK analysis set
Measure: Median (Full Range); unit: ng*min/mL
Arm/Group | Cohort 1: 6 ug/kg/Day Denileukin Diftitox | Cohort 2: 9 ug/kg/Day Denileukin Diftitox | Cohort 3: 12 ug/kg/Day Denileukin Diftitox
Number analyzed (Participants) | 3 | 5 | 2
ng*min/mL | 10300 [9860 to 12700] | 16900 [9980 to 21700] | 18600 [14000 to 23200]

6. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time 0 to Infinity (AUC(0-inf))
Description: Blood samples were collected before and 30 minutes after the start of infusion and immediately (0 minutes), 30, 60, 90, and 120 minutes after the end of infusion of denileukin diftitox. The samples were analyzed for the amount of denileukin diftitox in the serum using a validated ligand-binding assay with a LLOQ of 30 ng/mL. Serum PK data were analyzed using a non-compartmental analysis approach to obtain individual participant estimates of AUC(0-inf), which was then summarized as the median and full range for all participants and expressed as ng*min/mL.
Time Frame: Cycle 1 (Day 1)
Population: PK analysis set
Measure: Median (Full Range); unit: ng*min/mL
Arm/Group | Cohort 1: 6 ug/kg/Day Denileukin Diftitox | Cohort 2: 9 ug/kg/Day Denileukin Diftitox | Cohort 3: 12 ug/kg/Day Denileukin Diftitox
Number analyzed (Participants) | 3 | 4 | 1
ng*min/mL | 16800 [16300 to 18900] | 25200 [13300 to 28600] | 35600 [35600 to 35600]

7. Secondary Outcome: Terminal Phase Rate Constant (λz)
Description: Blood samples were collected before and 30 minutes after the start of infusion and immediately (0 minutes), 30, 60, 90, and 120 minutes after the end of infusion of denileukin diftitox. The samples were analyzed for the amount of denileukin diftitox in the serum using a validated ligand-binding assay with a LLOQ of 30 ng/mL. Serum PK data were analyzed using a non-compartmental analysis approach to obtain individual participant estimates of λz, which was then summarized as the median and full range for all participants and expressed in 1/minutes.
Time Frame: Cycle 1 (Day 1)
Population: PK analysis set
Measure: Median (Full Range); unit: 1/minutes
Arm/Group | Cohort 1: 6 ug/kg/Day Denileukin Diftitox | Cohort 2: 9 ug/kg/Day Denileukin Diftitox | Cohort 3: 12 ug/kg/Day Denileukin Diftitox
Number analyzed (Participants) | 3 | 4 | 1
1/minutes | 0.00746 [0.00647 to 0.00895] | 0.0103 [0.00656 to 0.0115] | 0.00793 [0.00793 to 0.00793]

8. Secondary Outcome: Terminal Elimination Phase Half-life (t1/2)
Description: Blood samples were collected before and 30 minutes after the start of infusion and immediately (0 minutes), 30, 60, 90, and 120 minutes after the end of infusion of denileukin diftitox. The samples were analyzed for the amount of denileukin diftitox in the serum using a validated ligand-binding assay with a LLOQ of 30 ng/mL. Serum PK data were analyzed using a non-compartmental analysis approach to obtain individual participant estimates of t1/2, which was then summarized as the median and full range for all participants and expressed in minutes.
Time Frame: Cycle 1 (Day 1)
Population: PK analysis set
Measure: Median (Full Range); unit: Minutes
Arm/Group | Cohort 1: 6 ug/kg/Day Denileukin Diftitox | Cohort 2: 9 ug/kg/Day Denileukin Diftitox | Cohort 3: 12 ug/kg/Day Denileukin Diftitox
Number analyzed (Participants) | 3 | 4 | 1
Minutes | 92.9 [77.5 to 107] | 67.8 [60.2 to 106] | 87.4 [87.4 to 87.4]

9. Secondary Outcome: Volume of Distribution at Terminal Phase (Vz)
Description: Blood samples were collected before and 30 minutes after the start of infusion and immediately (0 minutes), 30, 60, 90, and 120 minutes after the end of infusion of denileukin diftitox. The samples were analyzed for the amount of denileukin diftitox in the serum using a validated ligand-binding assay with a LLOQ of 30 ng/mL. Serum PK data were analyzed using a non-compartmental analysis approach to obtain individual participant estimates of Vz, which was then summarized as the median and full range for all participants and expressed as milliliters per kilogram (mL/kg).
Time Frame: Cycle 1 (Day 1)
Population: PK analysis set
Measure: Median (Full Range); unit: mL/kg
Arm/Group | Cohort 1: 6 ug/kg/Day Denileukin Diftitox | Cohort 2: 9 ug/kg/Day Denileukin Diftitox | Cohort 3: 12 ug/kg/Day Denileukin Diftitox
Number analyzed (Participants) | 3 | 4 | 1
mL/kg | 54.2 [46.8 to 57.3] | 45.2 [29.7 to 58.9] | 49.5 [49.5 to 49.5]

10. Secondary Outcome: Volume of Distribution at Steady State (Vss)
Description: Blood samples were collected before and 30 minutes after the start of infusion and immediately (0 minutes), 30, 60, 90, and 120 minutes after the end of infusion of denileukin diftitox. The samples were analyzed for the amount of denileukin diftitox in the serum using a validated ligand-binding assay with a LLOQ of 30 ng/mL. Serum PK data were analyzed using a non-compartmental analysis approach to obtain individual participant estimates of Vss, which was then summarized as the median and full range for all participants and expressed as mL/kg.
Time Frame: Cycle 1 (Day 1)
Population: PK analysis set
Measure: Median (Full Range); unit: mL/kg
Arm/Group | Cohort 1: 6 ug/kg/Day Denileukin Diftitox | Cohort 2: 9 ug/kg/Day Denileukin Diftitox | Cohort 3: 12 ug/kg/Day Denileukin Diftitox
Number analyzed (Participants) | 3 | 4 | 1
mL/kg | 59.8 [54.7 to 60.7] | 48.4 [32.3 to 62.3] | 54.1 [54.1 to 54.1]

11. Secondary Outcome: Total Clearance (CL)
Description: Blood samples were collected before and 30 minutes after the start of infusion and immediately (0 minutes), 30, 60, 90, and 120 minutes after the end of infusion of denileukin diftitox. The samples were analyzed for the amount of denileukin diftitox in the serum using a validated ligand-binding assay with a LLOQ of 30 ng/mL. SerumPK data were analyzed using a non-compartmental analysis approach to obtain individual participant estimates of CL, which was then summarized as the median and full range for all participants and expressed as milliliters/minutes/kilograms (mL/min/kg).
Time Frame: Cycle 1 (Day 1)
Population: PK analysis set
Measure: Median (Full Range); unit: mL/min/kg
Arm/Group | Cohort 1: 6 ug/kg/Day Denileukin Diftitox | Cohort 2: 9 ug/kg/Day Denileukin Diftitox | Cohort 3: 12 ug/kg/Day Denileukin Diftitox
Number analyzed (Participants) | 3 | 4 | 1
mL/min/kg | 0.404 [0.371 to 0.418] | 0.361 [0.321 to 0.679] | 0.393 [0.393 to 0.393]

12. Secondary Outcome: Recommended Dose
Description: This endpoint was combined with primary outcome measure, MTD
Time Frame: For each dose, first dose of study drug (Cycle 1 Day 1) to end of Cycle 1 (Day 21) (1 cycle = 3 weeks)
Population: This endpoint was combined with primary outcome measure, MTD
Groups:
- Denileukin Diftitox: Denileukin diftitox was IV-infused for 60 minutes (±10 minutes) daily from Day 1 through Day 5 of each Cycle (1 cycle = 3 weeks).
Arm/Group | Denileukin Diftitox
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From date of first dose up to 30 days after the last dose of study treatment, up to approximately 4 years 2 months
Description: Treatment-emergent adverse events and serious adverse events were reported. Adverse events were graded on a 5-point scale according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. The safety analysis set was used and included all participants who received at least one dose of study drug with at least one evaluable, post-baseline safety datum.
Arm/Group | Cohort 1: 6 ug/kg/Day Denileukin Diftitox | Cohort 2: 9 ug/kg/Day Denileukin Diftitox | Cohort 3: 12 ug/kg/Day Denileukin Diftitox
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/7 | 1/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/7 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: 6 ug/kg/Day Denileukin Diftitox (N=3) | Cohort 2: 9 ug/kg/Day Denileukin Diftitox (N=7) | Cohort 3: 12 ug/kg/Day Denileukin Diftitox (N=3)
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Aspartate Aminotransferase increased (Investigations) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hepatic Failure (Hepatobiliary disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: 6 ug/kg/Day Denileukin Diftitox (N=3) | Cohort 2: 9 ug/kg/Day Denileukin Diftitox (N=7) | Cohort 3: 12 ug/kg/Day Denileukin Diftitox (N=3)
Fatigue (General disorders) | 3 | 4 | 3
Pyrexia (General disorders) | 0 | 4 | 2
Oedema peripheral (General disorders) | 2 | 2 | 1
Malaise (General disorders) | 0 | 4 | 0
Face Oedema (General disorders) | 0 | 2 | 0
Generalised oedema (General disorders) | 0 | 1 | 1
Infusion site extravasation (General disorders) | 0 | 1 | 1
Injection site swelling (General disorders) | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 5 | 3
Aspartate aminotransferase increased (Investigations) | 2 | 5 | 3
Lymphocyte count decreased (Investigations) | 3 | 4 | 3
Platelet count decreased (Investigations) | 2 | 4 | 2
Lipase increased (Investigations) | 2 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 2 | 1
Neutrophil count decreased (Investigations) | 1 | 1 | 2
Weight increased (Investigations) | 1 | 1 | 2
Amylase increased (Investigations) | 1 | 1 | 1
Blood cholesterol increased (Investigations) | 1 | 2 | 0
White blood cell decreased (Investigations) | 1 | 1 | 1
Blood albumin decreased (Investigations) | 0 | 2 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Blood cholinesterase decreased (Investigations) | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0
Blood fibrinogen decreased (Investigations) | 0 | 0 | 1
Blood fibrinogen increased (Investigations) | 0 | 1 | 0
Cytomegalovirus test positive (Investigations) | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 4 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 5 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 4 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 3 | 3 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 4 | 3
Constipation (Gastrointestinal disorders) | 2 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 3
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Oral Herpes (Infections and infestations) | 0 | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 2 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 2
Capillary leak syndrome (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Conjunctival oedema (Eye disorders) | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0
Visual Impairment (Eye disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 2 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1
Antithrombin III deficiency (Congenital, familial and genetic disorders) | 0 | 0 | 1
Colour Blindness (Congenital, familial and genetic disorders) | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Central nervous system lesion (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other